CLINICAL TRIAL: NCT02446314
Title: A Randomized, Double-blind, Placebo-controlled Study Investigating the Effects of a Wild Blueberry Powder and a Wild Blueberry Extract on Cognition in Older Adults
Brief Title: An Investigation Into the Effects of a Wild Blueberry Powder and a Wild Blueberry Extract on Cognition in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Principal Investigator, Prof Claire Williams, Associate Professor in Behavioural Neuroscience, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RDG-001
Record Dates: First submitted 2015-04-27; First posted 2015-05-18 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-06

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator): Formulation containing inert artificially colored maltodextrin, once daily, in a 2-hard capsule regimen
  Interventions: Dietary Supplement: Placebo
- Wild Blueberry Powder - 450mg (Experimental): Formulation containing 225 mg wild blueberry powder + 22.5 mg L-Cysteine + 2.5 mg L-Glutathione + 250 mg placebo powder, once daily, in a 2-hard capsule regimen
  Interventions: Dietary Supplement: Wild Blueberry Powder - 450mg
- Wild Blueberry Powder - 900 mg (Experimental): Formulation containing containing 450 mg wild blueberry powder + 45 mg L-Cysteine + 5 mg L-Glutathione once daily, in a 2-hard capsule regimen
  Interventions: Dietary Supplement: Wild Blueberry Powder - 900 mg
- Wild Blueberry extract 100mg (Experimental): Formulation containing containing 100 mg wild blueberry powder + 10 mg L-Cysteine + 1 mg L-Glutathione + 389 mg of placebo, once daily, in a 2-hard capsule regimen
  Interventions: Dietary Supplement: Wild Blueberry extract 100mg

INTERVENTIONS:
Dietary Supplement: Placebo — Formulation containing inert artificially colored maltodextrin, once daily, in a 2-hard capsule regimen
  Arms: Placebo
Dietary Supplement: Wild Blueberry Powder - 450mg — Formulation containing 225 mg wild blueberry powder + 22.5 mg L-Cysteine @ 2.5 mg L-Glutathione 250 mg placebo powder, once daily, in a 2-hard capsule regimen
  Arms: Wild Blueberry Powder - 450mg
Dietary Supplement: Wild Blueberry Powder - 900 mg — Formulation containing 450 mg wild blueberry powder = 45 mg L-Cysteine + 5 mg L-Glutathione once daily, in a 2-hard capsule regimen
  Arms: Wild Blueberry Powder - 900 mg
Dietary Supplement: Wild Blueberry extract 100mg — Formulation containing 100 mg wild blueberry powder + 10 mg L-Cysteine + 1 mg L-Glutathione + 389 mg of placebo, once daily, in a 2-hard capsule regimen
  Arms: Wild Blueberry extract 100mg

SUMMARY:
The purpose of this study is to determine whether a 6 month dietary intervention with wild blueberry powder and extract stabilised with L-cysteine and L-glutathione have an effect on cognitive performance in participants aged between 65 - 80.

DETAILED DESCRIPTION:
Interventions: A placebo and two different wild blueberry products will be used in this study (see Table 1). A wild blueberry powder at two different doses and a single wild blueberry extract. The wild blueberry powder will be used at a 450 mg-dose, to which 45 mg of L-Cysteine and 5 mg of L-Glutathione will be added (wild blueberry powder-450), as well as at a 900 mg-dose, to which 90 mg of L-Cysteine and 10 mg of L-Glutathione will also be added (wild blueberry powder-900). The wild blueberry extract will consist of 100 mg of wild blueberry extract supplemented with 10 mg of L-Cysteine and 1 mg of L-Glutathione. Participants will be asked to consume two capsules daily with their normal breakfast. The capsules will be packed in blister packs with 4 capsules per blister. Each box contains 4 blisters (or a total of 16 capsules) in order to provide for 1 week of study medication, with 2 capsules remaining. Participants will be instructed to return the left-over investigational product weekly (i.e two capsules) using stamped addressed envelopes supplied by the experimenters. Weekly assessment of left-over investigational product will allow for continued compliance verification.

Procedure: The study comprises of a telephone screen and then six visits, including a familiarization visit (week T-1), three test visits (week 0, 12 and 24), and two control visits (week 6 and 18). Participants may stop the study treatment without stating any reason at any time during the study. In addition, a participant will be withdrawn from the study if: a subject requests discontinuation, he/she exhibits a serious adverse event to any component of the test product, the participant significantly violates the inclusion or exclusion criteria, an intercurrent illness emerges and/or the investigator's opinion is that withdrawal is appropriate and in the best interest of the participant. If a participant withdraws from the study, he/she will be encouraged to make a final visit as soon as possible, irrespective of the reason for withdrawal, to complete a final battery of cognitive tasks.

1. Screening: once a participant has indicated that they wish to join the trial they will be contacted by telephone for a brief screening session. The research associate (RA) will give a brief overview of the study and will ascertain that each interested volunteer is willing to participate for the entire duration of the study and to check that they fulfill our inclusion/exclusion criteria. Once confirmation of suitability for the study is confirmed, the RA will schedule their familiarization visit.
2. Familiarization Visit: Volunteers will be asked to attend the Nutritional Psychology Unit at the University of Reading where they will receive a detailed explanation on the study by the participating research associate and will be asked to sign the informed consent form before any study procedure starts. A log will be kept identifying all participants having signed the informed consent form (ICF) and the participant will be allocated a participant number. Once consent has been given, the inclusion/exclusion criteria will be checked once again and vital signs (blood pressure and heart rate) and anthropometric measurements (height, weight, BMI) will be taken. The participants will then be asked to complete a number of questionnaires and cognitive tasks comprising: (i) Yale Physical Activity Questionnaire; (ii) Frequency of Forgetting Questionnaire to give a baseline assessment of their memory performance; and (iii) Computerized Global Cognitive Health Assessments (NART, CERAD, MMSE, letter and category fluency; unless as a member of the Older Adult Panel these data have been collected from them in the preceding 3 months). Finally, participants will be given training on the cognitive test battery (tasks outlined below) that will be used during the study to reduce the chances of 'practice' adversely effecting performance on subsequent test days. Before leaving the laboratory, participants will be asked to keep a 72 hour food diary (consisting of 2 week days & 1 weekend day) so that background flavonoid intakes can be measured prior to the start of the intervention.
3. Test Visits (Weeks 0, 12 and 24): All of these sessions will be held in the morning (typically 8am-10am arrival time to suit participants individual needs). Participants will attend the laboratory in a fasted state and on arrival at the laboratory we will check participants still fulfill our inclusion/exclusion criteria, their general well-being, notification of any adverse events, any issues with compliance, and to check whether there have been changes to any concomitant medication. Blood pressure and heart rate will also be measured, and the food diary will be collected (week 0 and 24 only). They will then receive a standard low-flavonoid breakfast and will complete the battery of cognitive tasks (see below). Subjects will then be given their intervention (sufficient quantity until their next test session, in blister packs, weeks 0 and 12 only), and will then be requested to consume 2 capsules each day. At week 24 only, the Yale Physical Activity and Frequency of Forgetting questionnaires will also be administered, and weight will be measured.
4. Control Visits (weeks 6 & 18): These sessions can take place at any time of day to suit the participant. Participants will attend the laboratory at the University of Reading to collect the next 6 week supply of their intervention. During these visits we will check that participants still fulfill our inclusion/exclusion criteria, informally check their well-being, inquire whether there have been any adverse events, and confirm that there have not been any changes to their concomitant medication. At week 18 only participants will be given another copy of the 72 hour food diary (consisting of 2 week days & 1 weekend day and asked to complete this before they return for their test visit in week 24.

ELIGIBILITY:
Inclusion Criteria:

* Overall healthy volunteers as proven by medical history and/or physical examination and of all ethnicity and socioeconomic status
* Free-living
* Subjects with subjective memory complaints
* MMSE: 24-30
* Subjects are willing to maintain their normal eating habits and exercise habits to avoid changes in body weight over the duration of the study
* Being willing to complete the food diaries and questionnaires
* Able to give signed written informed consent
* Signed informed consent form

Exclusion Criteria:

* Use of complementary and alternative medicine
* History of metabolic disorder, diabetes, substance abuse
* Subjects diagnosed with psychiatric or neurological conditions
* Subjects using medications that might affect the outcome measures (such as antidepressant and sleeping medication), or planned changes

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire M Williams, PhD, Principal Investigator — University of Reaiding; Emilie Fromentin, PhD, Study Director — NATURIEX-DBS,, LLC
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Background] How, P.S., Ellis, J.A., Neshatdoust, S., Spencer, J.P.E. (2008). The impact of plant-derived flavonoids on mood, memory and motor skills in healthy older UK adults. Proceedings of the Nutrition Society, 67, E316.
- [Background] Krikorian R, Shidler MD, Nash TA, Kalt W, Vinqvist-Tymchuk MR, Shukitt-Hale B, Joseph JA. Blueberry supplementation improves memory in older adults. J Agric Food Chem. 2010 Apr 14;58(7):3996-4000. doi: 10.1021/jf9029332. PMID 20047325
- [Background] Macready AL, Kennedy OB, Ellis JA, Williams CM, Spencer JP, Butler LT. Flavonoids and cognitive function: a review of human randomized controlled trial studies and recommendations for future studies. Genes Nutr. 2009 Dec;4(4):227-42. doi: 10.1007/s12263-009-0135-4. Epub 2009 Aug 13. PMID 19680703
- [Background] Rendeiro C, Vauzour D, Kean RJ, Butler LT, Rattray M, Spencer JP, Williams CM. Blueberry supplementation induces spatial memory improvements and region-specific regulation of hippocampal BDNF mRNA expression in young rats. Psychopharmacology (Berl). 2012 Oct;223(3):319-30. doi: 10.1007/s00213-012-2719-8. Epub 2012 May 9. PMID 22569815
- [Background] Rendeiro C, Vauzour D, Rattray M, Waffo-Teguo P, Merillon JM, Butler LT, Williams CM, Spencer JP. Dietary levels of pure flavonoids improve spatial memory performance and increase hippocampal brain-derived neurotrophic factor. PLoS One. 2013 May 28;8(5):e63535. doi: 10.1371/journal.pone.0063535. Print 2013. PMID 23723987
- [Result] Whyte AR, Cheng N, Fromentin E, Williams CM. A Randomized, Double-Blinded, Placebo-Controlled Study to Compare the Safety and Efficacy of Low Dose Enhanced Wild Blueberry Powder and Wild Blueberry Extract (ThinkBlue) in Maintenance of Episodic and Working Memory in Older Adults. Nutrients. 2018 May 23;10(6):660. doi: 10.3390/nu10060660. PMID 29882843

RESULTS

PARTICIPANT FLOW:
Period: Zero to Twelve Weeks.
Arm/Group | Placebo | Wild Blueberry Powder - 450mg | Wild Blueberry Powder - 900 mg | Wild Blueberry Extract 100mg
Started | 30 | 30 | 31 | 31
Completed | 27 | 29 | 31 | 29
Not Completed | 3 | 1 | 0 | 2
Period: Thirteen to Twenty Four Weeks
Arm/Group | Placebo | Wild Blueberry Powder - 450mg | Wild Blueberry Powder - 900 mg | Wild Blueberry Extract 100mg
Started | 27 | 29 | 31 | 29
Completed | 27 | 28 | 29 | 28
Not Completed | 0 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Wild Blueberry Powder - 450mg | Wild Blueberry Powder - 900 mg | Wild Blueberry Extract 100mg | Total
Number analyzed (Participants) | 30 | 30 | 31 | 31 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (3.07) | 70.5 (2.87) | 70.3 (3.59) | 70.2 (4.30) | 70.5 (3.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 26 | 15 | 18 | 75
  Male | 14 | 4 | 16 | 13 | 47
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30 | 30 | 31 | 31 | 122

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Words Correctly Recognised.
Description: Participants indicate whether words presented on a monitor are from a list of 15 words previously presented auditorily (via headphones), or if they are novel foils.
Time Frame: 12, and 24 weeks
Measure: Mean (Standard Error); unit: proportion of words correctly recognised
Arm/Group | Placebo | Wild Blueberry Powder - 450mg | Wild Blueberry Powder - 900 mg | Wild Blueberry Extract 100mg
Number analyzed (Participants) | 27 | 28 | 29 | 28
proportion of words correctly recognised
  12 Weeks | 0.86 (0.02) | 0.85 (0.02) | 0.79 (0.02) | 0.90 (0.02)
  24 Weeks | 0.90 (0.02) | 0.88 (0.02) | 0.87 (0.02) | 0.88 (0.02)

2. Primary Outcome: Total Number of Correct Sequences Recalled
Description: Participants view an array of 9 white squares on a monitor which light up red in sequences of between 2 and 9. They are then required to press the correct squares in the sequence they were presented.
Time Frame: 12, and 24 weeks
Measure: Mean (Standard Error); unit: Correct number of sequences
Arm/Group | Placebo | Wild Blueberry Powder - 450mg | Wild Blueberry Powder - 900 mg | Wild Blueberry Extract 100mg
Number analyzed (Participants) | 27 | 28 | 29 | 28
Correct number of sequences
  12 Weeks | 15.15 (0.41) | 14.27 (0.40) | 15.42 (0.39) | 16.19 (0.39)
  24 Weeks | 15.56 (0.48) | 16.348 (0.47) | 15.921 (0.46) | 16.302 (0.46)

3. Primary Outcome: Combined Z Score of Delayed Words Recalled, Words Recognised, and Pictures Recognised.
Description: Combined Z score of proportion of words recalled, proportion of words recognised, and proportion of pictures recognised. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean. A negative change value reflects a decrease in memory or a worse outcome and a positive change value reflects an increase in memory or a better outcome
Time Frame: 12, and 24 weeks
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Placebo | Wild Blueberry Powder - 450mg | Wild Blueberry Powder - 900 mg | Wild Blueberry Extract 100mg
Number analyzed (Participants) | 27 | 28 | 29 | 28
z-score
  12 Weeks | 0.19 (0.11) | 0.08 (0.11) | 0.02 (0.11) | 0.28 (0.11)
  24 Weeks | 0.31 (0.09) | 0.13 (0.09) | 0.33 (0.08) | 0.2 (0.09)

4. Secondary Outcome: Combined Z Score of Mean Reaction Time Scores for Incongruent Attention Network and Stroop Task Trials.
Description: Combined Z Score of Mean Reaction Time Scores for Incongruent Attention Network and Stroop Task Trials. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean. A negative change value reflects a decrease in memory or a worse outcome and a positive change value reflects an increase in memory or a better outcome.
Time Frame: 12, and 24 weeks
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Placebo | Wild Blueberry Powder - 450mg | Wild Blueberry Powder - 900 mg | Wild Blueberry Extract 100mg
Number analyzed (Participants) | 27 | 28 | 29 | 28
z-score
  12 Weeks | 0.003 (0.067) | 0.009 (0.068) | -0.137 (0.064) | -0.037 (0.067)
  24 Weeks | -0.101 (0.065) | -0.176 (0.066) | -0.129 (0.062) | -0.075 (0.065)

5. Secondary Outcome: Combined Z Score of Proportion of Immediate Words Recalled, Number of Correct Serial 3 and Serial 7 Subtractions, Sternberg Task Coefficent of the Line
Description: Combined Z Score of Proportion of Immediate Words Recalled, Number of Correct Serial 3 and Serial 7 Subtractions, and the Coefficient of the Line for Reaction Time by Length of Sting During Probe Recall. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean. A negative change value reflects a decrease in memory or a worse outcome and a positive change value reflects an increase in memory or a better outcome
Time Frame: 12, and 24 weeks
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Placebo | Wild Blueberry Powder - 450mg | Wild Blueberry Powder - 900 mg | Wild Blueberry Extract 100mg
Number analyzed (Participants) | 27 | 28 | 29 | 28
z-score
  12 Weeks | 0.12 (0.09) | -0.03 (0.08) | -0.13 (0.08) | 0.03 (0.08)
  24 Weeks | 0.1 (0.07) | -0.01 (0.07) | -0.04 (0.07) | 0.02 (0.07)

6. Secondary Outcome: Systolic Blood Pressure
Description: LMM analysis of intervention group x 12 and 24 wk test session. Baseline blood pressure entered as a covariate.
Time Frame: 12, and 24 weeks.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Wild Blueberry Powder - 450mg | Wild Blueberry Powder - 900 mg | Wild Blueberry Extract 100mg
Number analyzed (Participants) | 27 | 28 | 29 | 28
mmHg
  12 Weeks | 124.11 (2.09) | 124.51 (2.05) | 125.16 (2.03) | 118.62 (2.15)
  24 Weeks | 119.63 (2.05) | 122.39 (2.01) | 119.79 (1.99) | 114.72 (2.11)
Statistical Analysis 1: Comparison: Placebo vs Wild Blueberry Powder - 450mg vs Wild Blueberry Powder - 900 mg vs Wild Blueberry Extract 100mg; Test type: Superiority; p = .04, Linear Mixed Model / Baseline Covariate

7. Secondary Outcome: Diastolic Blood Pressure
Description: LMM analysis of intervention group x 12 and 24 wk test session. Baseline blood pressure entered as a covariate.
Time Frame: 12, and 24 weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Wild Blueberry Powder - 450mg | Wild Blueberry Powder - 900 mg | Wild Blueberry Extract 100mg
Number analyzed (Participants) | 27 | 28 | 29 | 28
mmHg
  12 Weeks | 72.70 (1.16) | 74.85 (1.13) | 72.30 (1.09) | 72.30 (1.13)
  24 Weeks | 71.71 (1.21) | 73.54 (1.18) | 71.23 (1.13) | 71.45 (1.17)
Statistical Analysis 1: Comparison: Placebo vs Wild Blueberry Powder - 450mg vs Wild Blueberry Powder - 900 mg vs Wild Blueberry Extract 100mg; Test type: Superiority; p > .05, Linear Mixed Model / Baseline Covariate

8. Secondary Outcome: Heart Rate
Description: LMM analysis of intervention group x 12 and 24 wk test session. Baseline heart rate entered as a covariate.
Time Frame: 12, and 24 weeks.
Measure: Mean (Standard Error); unit: beats/min
Arm/Group | Placebo | Wild Blueberry Powder - 450mg | Wild Blueberry Powder - 900 mg | Wild Blueberry Extract 100mg
Number analyzed (Participants) | 27 | 28 | 29 | 28
beats/min
  12 Weeks | 68.33 (1.02) | 69.16 (0.98) | 66.07 (0.95) | 67.56 (0.99)
  24 Weeks | 68.62 (1.22) | 67.47 (1.18) | 67.11 (1.15) | 70.04 (1.19)
Statistical Analysis 1: Comparison: Placebo vs Wild Blueberry Powder - 450mg vs Wild Blueberry Powder - 900 mg vs Wild Blueberry Extract 100mg; Test type: Superiority; p > .05, Linear Mixed Model / Baseline Covariate

9. Secondary Outcome: Positive Affect Score
Description: As measured by the positive mood scale derived from the Positive and Negative Affect Schedule. This measure consists of 10 words relating to positive affect. The participants is asked to rate how they feel about each word from 1 (very slightly/not at all) to 5 (extremely) with a minimum score of 5 and maximum of 50. A higher score relates to higher positive affect.
Time Frame: 12, and 24 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Wild Blueberry Powder - 450mg | Wild Blueberry Powder - 900 mg | Wild Blueberry Extract 100mg
Number analyzed (Participants) | 27 | 28 | 29 | 28
units on a scale
  12 Weeks | 31.29 (0.92) | 31.18 (0.90) | 32.10 (0.92) | 31.30 (0.92)
  24 Weeks | 31.06 (0.84) | 31.07 (0.82) | 30.83 (0.83) | 31.96 (0.83)
Statistical Analysis 1: Comparison: Placebo vs Wild Blueberry Powder - 450mg vs Wild Blueberry Powder - 900 mg vs Wild Blueberry Extract 100mg; Test type: Superiority; p > .05, Linear Mixed Model / Baseline Covariate

10. Secondary Outcome: Negative Affect Score
Description: As measured by the negative mood scale derived from the Positive and Negative Affect Schedule. This measure consists of 10 words relating to negative affect. The participants is asked to rate how they feel about each word from 1 (very slightly/not at all) to 5 (extremely) with a minimum score of 5 and maximum of 50. A higher score relates to higher negative affect.
Time Frame: 12, and 24 weeks.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Wild Blueberry Powder - 450mg | Wild Blueberry Powder - 900 mg | Wild Blueberry Extract 100mg
Number analyzed (Participants) | 27 | 28 | 29 | 28
units on a scale
  12 Weeks | 12.04 (0.44) | 13.14 (0.42) | 11.72 (0.42) | 11.53 (0.44)
  24 Weeks | 12.17 (0.41) | 12.18 (0.40) | 12.11 (0.40) | 11.57 (0.41)
Statistical Analysis 1: Comparison: Placebo vs Wild Blueberry Powder - 450mg vs Wild Blueberry Powder - 900 mg vs Wild Blueberry Extract 100mg; Test type: Superiority; p > .05, Linear Mixed Model / Baseline Covariate

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Wild Blueberry Powder - 500mg: Wild Blueberry Powder - 450mg: Formulation containing 225 mg wild blueberry powder + 45 mg L-Cysteine + 5 mg L-Glutathione + 250 mg placebo powder, once daily, in a 2-hard capsule regimen
- Wild Blueberry Powder - 1000 mg: Wild Blueberry Powder - 1000 mg: Formulation containing 900 mg wild blueberry powder + 90 mg L-Cysteine + 10 mg L-Glutathione once daily, in a 2-hard capsule regimen
- Wild Blueberry Extract 111mg: Wild Blueberry extract 100mg: Formulation containing 100 mg wild blueberry powder + 10 mg L-Cysteine + 1 mg L-Glutathione + 889 mg of placebo, once daily, in a 2-hard capsule regimen
Arm/Group | Placebo | Wild Blueberry Powder - 500mg | Wild Blueberry Powder - 1000 mg | Wild Blueberry Extract 111mg
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 1/30 | 0/30 | 1/31 | 2/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Wild Blueberry Powder - 500mg (N=30) | Wild Blueberry Powder - 1000 mg (N=31) | Wild Blueberry Extract 111mg (N=31)
Diarrhoea / Looser Stool (Gastrointestinal disorders) | 1 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No